CLINICAL TRIAL: NCT05290155
Title: The Safety and Clinical Efficacy of Human CD7 CAR-T Cell Therapy for Patients With Relapsed/Refractory CD7 Positive T Cell Hematological Maliganacies
Brief Title: Anti-CD7 CAR-T Cell Therapy for Relapse and Refractory CD7 Positive T Cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, principal investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHYSXY-202105-CD7-CART
Record Dates: First submitted 2022-03-09; First posted 2022-03-22 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma; T-cell Acute Lymphoblastic Leukemia; Peripheral T Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: chimeric antigen receptor T cell; T lymphoblastic lymphoma/leukemia; T cell non-Hodgkin lymphoma; CD7
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Leukemia; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD7 CAR T cells (Experimental): Administration with anti-CD7 CAR-T cells in the relapsed/refractory T cell hematological malignancy patients
  Interventions: Drug: anti-CD7 CAR-T cells

INTERVENTIONS:
Drug: anti-CD7 CAR-T cells — Administration with anti-CD7 CAR-T cells in the relapsed/refractory T cell hematological malignancy patients

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CAR T cell treatment targeting CD7 in patients with relapsed or refractory CD7 positive T-cell hematological maliganacies

DETAILED DESCRIPTION:
This study is single-armed，open lable，dose escalation clinical trial.The main purpose is to evaluate the safety and efficacy of anti-CD7 CAR-T cells in relapsed/refractory patients with CD7 positive T cell malignancies,including T lymphoblastic lymphoma/leukemia ,T-cell non-Hodgkin lymphoma(peripheral T cell lymphoma,NOS,angioimmunoblastic T cell lymphoma and anaplastic large cell lymphoma).There will be three CAR T cell dose groups:0.25*10^6 cells per kilogram of body weight;0.5*10^6 cells per kilogram of body weight，1 *10^6 ells per kilogram of body weight.

ELIGIBILITY:
Inclusion criteria

1. Fourteen to 70 Years Old, Male and female;
2. Expected survival > 12 weeks; ECOG score 0-2;
3. Confirmed diagnosis of acute T cell leukemia and screened for CD7 positive,including following conditions:a. Patients who do not get a CR with ≥2 prior induction therapy b. Those who achieves CR, but have a early relapse(<12months),or a late relapse (>=12months) failing to acheive a CR after re-induction chemotherapy c. For any Patiens failed ASCT/allo-SCT
4. Relapsed and refractory patients with diagnosis of CD7 positive T cell lymphoma have had≥2 prior lines of therapy,who do not acheive at least a PR, or have a relapse including:a. Peripheral T cell lymphoma NOS, or b.Angioimmunoblastic T cell lymphoma,or c. Anaplastic large cell lymphoma c.Disease can be assessed(BM or CT scan)
5. Confirmed T lymphoblastic lymphoma：a. Patients who do not get a PR with ≥2 induction chemotherapy or a CR with ≥ 4 induction chemotherapy b. Relapsed patients failing to achieve a CR after 1 line salvage chemotherapy c. For any Patients failed ASCT/allo-SCT .Disease can be assessed(BM or CT scan)
6. The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators;
7. Liver, kidney and cardiopulmonary functions meet the following requirements: a. Ccr≥60mL/min(Cockcroft Gault) b. Left ventricular ejection fraction >50%; c.Baseline oxygen saturation>92%; d. Total bilirubin ≤ 1.5×ULN; e. ALT and AST≤ 3×ULN;
8. Able to understand and sign the Informed Consent

Exclusion Criteria:

1. Malignant tumors other than T cell malignancies within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
2. Uncontrolled infection including bacteral or virus or fugal disease;patients with positive HBsAg or HBcAb and positive peripheral blood HBV DNA titer detection ;HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; syphilis positive;
3. Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening),myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia,liver, kidney, or metabolic disease;
4. Any uncontrolled disease may affect entry
5. Current or history of CNS involvement by malignancy.Known history or presence of clinically relevant central nervous system (CNS) pathology.Patients with a known history or prior diagnosis other immunologic or inflammatory disease affecting the CNS (such as epilepsy)
6. Patients who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
7. Subjects treated with anti-PD1 or anti-PDL1 therapies within 3months before enrollment
8. Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pr egnancy within 1 year after cell transfusion;
9. Active or uncontrollable infection requiring systemic therapy Received CAR-T treatment or other gene therapies before enrollment;
10. Kown be allergic to anti-TRBC1 CAR-T cells or drugs(Fludarabine or Cyclophophamide)
11. The investigators consider other conditions unsuitable for enrollment.
12. Patients who may not be able to sign the Informed Consent due to disease,or who do not understand or unwillingness or inability to comply with research requirements

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days post infusion
  The occurence of study related adverse effects defined by NCI CTCAE5.0

SECONDARY OUTCOMES:
CAR-T cell expansion | 2 years post infusion
  Using flow cytometry to reveal cell surface expression of the CAR protein on T cells;and using quantitative polymerase chain reaction to detect DNA copies of the transgene irrespective of gene expression(per ug DNA) to evaluate anti-CD7 CAR-T cell expansion after infusion
CAR-T cell persistence | 2 years post infusion
  Using flow cytometry to reveal cell surface expression of the CAR protein on T cells;and using quantitative polymerase chain reaction to detect DNA copies of the transgene irrespective of gene expression(per ug DNA) to evaluate anti-CD7 CAR-T cell persistence after infusion
Number of CD7+ lymphocytes of peripheral blood | 2 years post infusion
  To evaluate CD7 positive cells of peripheral blood after infusion
Total response rate (ORR) after administration | 3 months post infusion
  CR+CRi for T-ALL ;CR+PR for T cell lyphoma and T lymphoblastic lymphoma
Duration of remission (DOR) after administration | 2 years post infusion
  Duration of remission (DOR) after administration
Overall survival(OS) after administration | 2 years post infusion
  Overall Survival (OS)after administration
Progression Free Survival (PFS) after administration | 2 years post infusion
  Progression Free Survival (PFS) after administration

OTHER OUTCOMES:
Immunogenicity of CAR-T cells | 2 years post infusion
  Using flow cytometry to detect whether anti-car antibodies are contained in serum of patients receiving CAR-T cells infusion,and to evaluate the number of participants with antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin G Song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xianmin General Song, Shanghai, China

IPD SHARING:
Plan to Share IPD: No